CLINICAL TRIAL: NCT01601860
Title: Evaluation of Maternal and Perinatal Outcomes Associated With the Use of Non-pharmacological in Parturients in Active Phase of Labor
Brief Title: The Maternal and Perinatal Outcomes Associated With the Use of Non-pharmacological in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alessandra Cristina Marcolin, Prof. Dra., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR444841
Record Dates: First submitted 2011-09-19; First posted 2012-05-18 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Pain
Keywords: Labor; vaginal delivery; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Active Comparator: Control Group Pregnant women who receive assistance from the routine CRSM MATER care, not being assisted by the physiotherapist, but that will be evaluated at the same time in the intervention group.
  Interventions: Other: Other: Routine care
- Intervention Group (Experimental): Experimental: Intervention Group Pregnant women who receive the application the combination of non-pharmacological resources according to cervical dilation: Walking (with cervical dilation between 4 and 5 cm) Alternating stance associated with ENT (cervical dilatation from 6 to 7 cm) Shower (with dilation> 7 cm);
  Interventions: Other: Use of non-pharmacological

INTERVENTIONS:
Other: Use of non-pharmacological — Other: Non-pharmacological resources
  A sequence of non-pharmacological resources were applied to the patient by the researcher according to uterine cervical dilation, as follows:
  * Walking (with cervical dilation between 4 and 5 cm)
  * Alternating stance associated with ENT (cervical dilatation from 6 to 7 cm)
  * Shower (with dilation> 7 cm);
  Arms: Intervention Group
Other: Other: Routine care — Other: Routine care Routine care of the institution performed by the staff, without the presence of the researcher that included offering a balanced meal, continuous support with the presence of a partner or family throughout labor, use of oxytocin when prescribed by the staff, use of drug analgesia when requested by the patient.
  Arms: Control

SUMMARY:
Although there are studies that investigated the use of non-pharmacological pain relief and correction of dystocia during labor, there are few randomized controlled trials, especially related to combined protocols that use such resources. The use of combined protocols could potentiate the effects of resource use alone, evidencing the need for more studies related to the topic, as well as the effects of these methods on maternal and perinatal outcomes. In order to verify the effect of these methods in various stages of labor, childbirth and immediately becomes necessary to conduct a randomized controlled trial well-designed and adequate sample size that can make the future systematic reviews that can definitely conclude about the potential effectiveness of protocols that use combined resources to non-pharmacological pain relief in labor. Aim of our study is to evaluate the effects of a protocol of non-pharmacological resources on pain of pregnant women in the active phase of cervical dilatation and compared with controls.

DETAILED DESCRIPTION:
Labor is a natural physiologic process triggered by mechanical and hormonal events that promote uterine contractions. Several non-pharmacological resources can be used during labor, such as relaxation techniques and ongoing support, maternal mobility, walking, breathing exercises, massage, Swiss ball, stool, shower, whirlpool and application of transcutaneous electrical stimulation (ENT .) Despite the role of physiotherapy in labor is not an established practice in public hospitals, it is expected that with the evidence of the benefits of non-pharmacological resources at this time, managers and health professionals validate the importance of interdisciplinary care in pregnancy - postpartum. The aim of this study is to evaluate the effects of resources on non-pharmacological pain of mothers in the active phase of cervical dilatation when compared to controls. This research is a randomized, controlled clinical study that includes pregnant women randomly assigned to two groups: Intervention Group (IG) women who will use the following sequence features: ambulation (with cervical dilatation of 4 to 5 cm), alternating stance associated with ENT (cervical dilatation from 6 to 7 cm) and a shower (with dilation> 7 cm) for 40 minutes each resource; Control Group (CG) women who will not use any physical therapy resource, are subject only to routine procedures of maternity care . For pain assessment will use the Visual Analogue Scale - VAS and the body diagram of the location and spatial distribution of pain. Results are presented in tables and graphs made to better understand the comparisons between the control and intervention. To compare maternal morbidity, obstetric and neonatal between groups will be used Fisher's exact test or chi-square.

ELIGIBILITY:
Inclusion Criteria:

* Agreement of the patient to participate in the study after reading and signing the consent form;

  * primigravida;
  * Pregnancy unique;
  * Gestational age> 37 weeks;
  * fetal cephalic presentation;
  * chorioamniotic intact membranes;
  * spontaneous labor;
  * Admission to the beginning of the active phase of dilatation (4 cm cervical dilatation);
  * Dynamics between 2 and 4 uterine contractions in ten minutes;
  * Lack of maternal and fetal pathologies;
  * literate;
  * Absence of cognitive problems.

Exclusion Criteria:

Intolerance to non-pharmacological application of resources;

* Increased pain by the woman that prevents the completion of the intervention;
* Want to stop the intervention;
* Suspected acute suffering;
* Indication of cesarean section.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra C Marcolin, Professor, Principal Investigator — Faculty of Medicine of São Paulo University
Locations (1):
- Professor, Department of Gynecology and Obstetrics, Faculty of Medicine of Ribeirão Preto, University of São Paulo., Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Frenea S, Chirossel C, Rodriguez R, Baguet JP, Racinet C, Payen JF. The effects of prolonged ambulation on labor with epidural analgesia. Anesth Analg. 2004 Jan;98(1):224-229. doi: 10.1213/01.ANE.0000090317.01876.D9. PMID 14693624

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Experimental: Intervention Group Pregnant women who receive the application the combination of non-pharmacological resources according to cervical dilation: Walking (with cervical dilation between 4 and 5 cm) Alternating stance associated with ENT (cervical dilatation from 6 to 7 cm) Shower (with dilation> 7 cm);
  Use of non-pharmacological: Other: Non-pharmacological resources
  A sequence of non-pharmacological resources were applied to the patient by the researcher according to uterine cervical dilation, as follows:
  * Walking (with cervical dilation between 4 and 5 cm)
  * Alternating stance associated with ENT (cervical dilatation from 6 to 7 cm)
  * Shower (with dilation> 7 cm);
Period: Overall Study
Arm/Group | Intervention Group | Control
Started | 40 | 40
Completed | 19 | 31
Not Completed | 21 | 9

BASELINE CHARACTERISTICS:
Population: Low-risk primigravidae women admitted to the maternity ward in the active phase of labor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 21.8 (4.22) | 22 (4.49) | 21.9 (4.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Low-risk primigravidae women admitted to the maternity ward in the active phase of labor.
  Participants
    Female | 40 | 40 | 80
    Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: Kilograms per square meter] | 28.4 (5.36) | 28.6 (4.94) | 28.5 (5.15)
School degree [Count of Participants; unit: Participants]
  Elementary school | 13 | 9 | 22
  Middle school | 24 | 27 | 51
  High school | 3 | 4 | 7
Marital status [Count of Participants; unit: Participants]
  Single | 6 | 13 | 19
  Married | 11 | 8 | 19
  with partner | 23 | 19 | 42
Paid employment, [Count of Participants; unit: Participants] | 17 | 12 | 29
PPW (pre-pregnancy weight) [Mean (Standard Deviation); unit: Kilograms per square meter] | 60.5 (13) | 61.1 (14.4) | 60.8 (13.7)
PDW (pre-delivery weight) [Mean (Standard Deviation); unit: Kilograms per square meter] | 72.6 (14.7) | 73.6 (14.4) | 73.1 (14.5)
Height [Mean (Standard Deviation); unit: centimeters] | 1.6 (0.07) | 1.6 (0.05) | 1.6 (0.06)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Requested Analgesia During the Active Phase of Childbirth
Description: Average uterine cervical dilation of the patient who requested analgesia for pain relief. Data captured from the medical record by the partograph.
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Active Comparator: Control Group Pregnant women who receive assistance from the routine CRSM MATER care, not being assisted by the physiotherapist, but that will be evaluated at the same time in the intervention group.
  Other: Routine care: Other: Routine care Routine care of the institution performed by the staff, without the presence of the researcher that included offering a balanced meal, continuous support with the presence of a partner or family throughout labor, use of oxytocin when prescribed by the staff, use of drug analgesia when requested by the patient.
- Intervention Group: Experimental: Intervention Group Pregnant women who receive the application the combination of non-pharmacological resources according to cervical dilation: Walking (with cervical dilation between 4 and 5 cm) Alternating stance associated with ENT (cervical dilatation from 6 to 7 cm) Shower (with dilation> 7 cm);
  Use of non-pharmacological: Other: Non-pharmacological resources
  A sequence of non-pharmacological resources were applied to the patient by the researcher according to uterine cervical dilation, as follows:
  * Walking (with cervical dilation between 4 and 5 cm)
  * Alternating stance associated with ENT (cervical dilatation from 6 to 7 cm)
  * Shower (with dilation> 7 cm).
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 37 | 35

2. Primary Outcome: The Moment in Centimeters That Women Requested Analgesia During the Active Phase of Childbirth, Analyzed by Cevical Dilation.
Description: Moment when a patient requested analgesia for pain relief. Data captured from the medical record by the partograph.
  A partogram was used, which is a printed document and allows the registration of all procedures and complications that occurred during labor, showing the conditions of the parturient and the fetus during this phase. This information is noted on a graph that makes it possible to assess all labor and duration. The doctor filled out the partograph and assessed the patient during labor, and she did not know which group belonged to the patient
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Groups:
- Control: The moment in centimeters that women requested analgesia during the active phase of childbirth, analyzed by cevical dilation.
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  4- 5 cm | 19 | 1
  6 - 7 cm | 16 | 8
  > 7 cm | 2 | 26
  Did not receive analgesia | 3 | 5

3. Primary Outcome: Average Duration of the Expulsive Period When Compared to Groups
Description: Assess the duration of the expulsion period and compare between groups
Time Frame: Starts with 10 centimeters of dilation until delivery
Population: [Not Specified]
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
minutes | 26 [7 to 135] | 18.5 [5 to 140]

4. Primary Outcome: Types of Dystocia (Functional, Secondary Stop of Dilation and Fetal Offspring) Between Groups
Description: Analyze and compare between the groups the types of dystocia.
  Dystocia:
  b.1) Functional dystocia was considered when cervical dilation increased progressively, but with a speed less than 1 centimeter per hour; b.2) Secondary stop of the dilation was considered when there were 2 vaginal touches with the same cervical dilation in an interval of at least two hours, without being total.
  b.3) Secondary descent stop was considered when, with complete dilation of the uterine cervix, the same height of fetal descent was found in two successive touches with an interval of one hour (Protocol Royal College of Obstetricians and Gynecologists, 2012).
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  functional | 24 | 17
  secondary stop of dilation | 6 | 3
  Secondary descent stop | 4 | 6
  without dystocia | 6 | 14

5. Primary Outcome: Admission Numbers to a Neonatal Intensive Care Unit Between Groups.
Description: Consider and compare neonatal admission to an intensive care unit between groups, attracted by the partogram
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 34 | 26

6. Primary Outcome: Number of Newborns With Apgar Scores of 1 and 5 Minutes, Less Than or Greater Than 7.
Description: Analyze and compare Apgar scores of the 1-min >7 and 5-min >7, between groups. The APGAR score reflects the degree of fetal maturity and predicts healthy child development. It is a scale that can vary from 0 to 10, which 0 is a bad vitality and 10 is an excellent score. When the APGAR score is below 7, especially in the fifth minute, it is a warning sign to give special attention to the newborn.
  Newborns who have an Apgar in the first minute greater than 7, demonstrate good birth conditions.
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  1-min >7 | 31 | 30
  5-min >7 | 40 | 40

7. Primary Outcome: Frequency of Suspected Fetal Distress, Between Groups
Description: Evaluate the frequency of suspected fetal distress with the presence of meconium release.
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 2 | 1

8. Secondary Outcome: Moment of Rupture of the Chorioamniorex Between the Groups.
Description: Observe if the groups had different types of cervical obstetric dilatation when a chorioamniorexis occurred.
Time Frame: 10 hours
Population: [Not Specified]
Measure: Median (95% Confidence Interval); unit: centimeters
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
centimeters | 7 [5 to 10] | 8 [6 to 10]

9. Secondary Outcome: Incidence in the Type of Delivery (Cesarean Section, Normal Delivery With Laceration, Episiotomy, Forceps and Normal Delivery).
Description: Type of delivery (cesarean section, normal delivery with laceration, episiotomy, forceps and normal delivery), collected by the partograph found in the medical record.
Time Frame: 10 hours
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  Cesarean section | 10 | 6
  normal birth | 3 | 8
  childbirth forcep | 4 | 1
  delivery with episiotomy | 17 | 14
  delivery with laceration | 6 | 11

10. Secondary Outcome: Number of Puerperal Women Who Present Hemorrhage in the Immediate Puerperium With Hemodynamic Repercussions Between Groups.
Description: Evaluate and compare the presence of hemorrhage with hemodynamic repercussions between groups (requiring surgical approach and / or blood transfusion)
Time Frame: immediately postpartum up to 2 days after childbirth
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 2 | 0

11. Secondary Outcome: The Number of Puerperal Infections Between Groups.
Description: Analyze and compare between the groups the number of puerperal infection
Time Frame: immediately postpartum up to 2 days after childbirth
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: [Not specified]
Description: Postpartum complication (Hemorrhage)
Arm/Group | Intervention Group | Control
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=40) | Control (N=40)
Postpartum complication (Hemorrhage) * [1] (Pregnancy, puerperium and perinatal conditions) | 0 | 2

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No